CLINICAL TRIAL: NCT05381792
Title: A Pilot Study to Assess Serial Gut Microbiome and a Panel of Bacterial Gene Markers (M3) Changes After Endoscopic Resection of Colorectal Advanced Neoplasia
Brief Title: Serial Gut Microbiome and Bacterial Gene Markers Changes After Endoscopic Resection of Colorectal Advanced Neoplasia
Acronym: M3-CAN
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Louis Ho Shing Lau, Assistant Professor (clinical), Chinese University of Hong Kong
Other Study IDs: 2022.127
Record Dates: First submitted 2022-05-12; First posted 2022-05-19 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Colorectal Cancer; Colorectal Neoplasms; Colorectal Adenoma
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Known colorectal advanced neoplasia group: Subjects with known colorectal advanced neoplasia and requiring endoscopic resection
  Interventions: Diagnostic Test: Bacterial gene markers test

INTERVENTIONS:
Diagnostic Test: Bacterial gene markers test — Bacterial gene markers test using qPCR

SUMMARY:
The investigators hypothesize that gut microbiome composition and the four bacterial gene markers (M3) show dynamic changes after endoscopic resection of advanced neoplasia, some key bacteria are associated with restoration of gut microbiome after endoscopic resection.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is one of the most common cancers in Hong Kong with more than 5,500 new cases annually. The majority of CRC cases are derived from benign colorectal adenomas through the process of adenoma-carcinoma sequence. Since this process takes several years, early detection and endoscopic resection of colorectal adenomas are important to reduce the incidence and mortality of CRC. Currently, colonoscopy is the gold standard for detection for colorectal adenomas. Endoscopic resection including endoscopic submucosal dissection (ESD) and endoscopic mucosal resection (EMR) can serve as minimally invasive treatment options for colorectal neoplasia. Compared with EMR, due to the general association with higher rates of en bloc, R0, and curative resections and a lower rate of local recurrence, ESD is an established and effective treatment modality for advanced adenoma (AA) and early-stage CRC.

Increasing studies showed a close crosstalk between the gut microbiome and colorectal neoplasia. Altered microbiome environment is associated with the initiation and progression of CRC and its precancerous lesions. Most studies focused on the gut microbiota changes in individuals with CRC and adenomas, and the potential microbial role in the progression of colorectal neoplasia. Conversely, the potential influence of CRC or adenomas on the gut microbiota is unclear. Only one study has depicted microbiota changes after the endoscopic removal of colorectal adenomas with limited follow up timepoints. Due to a high rate of recurrence of colorectal adenomas after endoscopic removal, surveillance colonoscopy is required depending on the size, number, and histology of polyps in the index coloscopy. Apart from these risk factors, reestablishment of gut microbiome after polyp resection may also play a role in the recurrence of adenomas.

Recently, a panel of bacterial gene markers including "m3" from Lachnoclostridium, Fusobacterium nucleatum (Fn), Bacteroides clarus (Bc) and Clostridium hathewayi (Ch) showed high diagnostic accuracy for CRC (82.3%) and adenomas (64.2%). The combination of these four bacterial gene markers (known as M3) has also been proven to be useful in detecting adenoma recurrence after polypectomy in a retrospective study. However, how these bacteria markers change after polypectomy and whether there are some associations between changes of bacteria gene markers and post resection restoration of the gut microbiome remain unclear.

This pilot study aims to determine serial gut microbiome composition changes, and changes in levels of the panel of four bacterial gene markers (M3) after endoscopic resection of colorectal advanced neoplasia, and factors associated with restoration of gut microbiome composition after endoscopic resection.

ELIGIBILITY:
Inclusion Criteria:

* Subjects require endoscopic resection (e.g. endoscopic mucosal resection or endoscopic submucosal dissection) for advanced adenoma or early-stage colorectal cancer;
* Aged 18-90 years old;
* Written informed consent obtained.

Exclusion Criteria:

* Absolute contraindications to colonoscopy (e.g. perforation, intestinal obstruction, unstable cardiopulmonary status);
* Contraindications to endoscopic resection (e.g. active gastrointestinal bleeding, uninterrupted anticoagulation or dual antiplatelets);
* Known pregnancy or lactation;
* Advanced comorbid conditions (defined as American Society of Anesthesiologists grade 4 or above);

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with known colorectal advanced neoplasia
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Serial bacterial gene markers changes (Fn, m3, Bc and Ch) after endoscopic resection of colorectal advanced neoplasia. | 6 months
  Bacterial gene markers change tested by quantitative polymerase chain reaction (qPCR)
Serial gut microbiome changes after endoscopic resection of colorectal advanced neoplasia. | 6 months
  Gut microbiome change tested by metagenomic sequencing

SECONDARY OUTCOMES:
The differences in the bacterial gene markers (Fn, m3, Bc and Ch) between different sites/sizes/pathology of advanced adenoma | 6 months
  Bacterial gene markers tested by qPCR
The differences in the bacterial gene markers (Fn, m3, Bc and Ch) between different stages of CRC | 6 months
  Bacterial gene markers tested by qPCR
The differences in the bacterial gene markers (Fn, m3, Bc and Ch) between advanced adenoma and CRC | 6 months
  Bacterial gene markers tested by qPCR

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Shatin, New Territories, Hong Kong

IPD SHARING:
Plan to Share IPD: No